CLINICAL TRIAL: NCT04027634
Title: Feasibility and Preliminary Effect of Baduanjin Program for People Diagnosed With Schizophrenia: A Pilot Randomized Controlled Trial
Brief Title: Feasibility and Preliminary Effect of Baduanjin Program for People Diagnosed With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chiu-Yueh Yang, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: JIRB12-S-019
Record Dates: First submitted 2019-07-13; First posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Randomized Controlled Trial
Keywords: Baduanjin program; body mass index; metabolic parameters; schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: The participants were divided into experimental and control groups through block randomization.
Who Masked: Participant
Masking Description: The data of the five metabolic indexes, height, and BW were collected by a research assistant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group (CG) received routine care and was required to walk during 6-7 pm.
- Baduanjin program (Experimental): The entire program continued for 3 months (mid-September to mid-December 2014), and the intervention was performed for 60 min 3 times per week; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Interventions: Other: Baduanjin program

INTERVENTIONS:
Other: Baduanjin program — This exercise program aimed to increase patient participation and control their BW through Baduanjin program. The entire program continued for 3 months (mid-September to mid-December 2014), and the intervention was performed for 60 min 3 times per week; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Arms: Baduanjin program

SUMMARY:
Introduction Low levels of physical activity and central obesity contribute to metabolic syndrome in patients with schizophrenia.

Aim This study was to examine the effectiveness of Baduanjin program on body mass index (BMI) and five metabolic parameters in participants with chronic schizophrenia.

Methods A randomized controlled trial was conducted in a psychiatric center in northern Taiwan. The eligibility criteria included BMI > 25 kg/m2, or with metabolic syndrome. Twenty-two participants were randomized to two groups using blocked randomization. The experimental group was provided with an 8-session Baduanjin program for 12 weeks (1 h, thrice times per week), while the control group received routine care.

DETAILED DESCRIPTION:
This study was conducted in a large psychiatric center that has 10 residential rehabilitation units. Residents were allowed to walk for 20 min during 6-7 pm every day, and each unit could accommodate approximately 50 residents. In this study, patients on the schizophrenia spectrum were invited to receive screening for metabolic syndrome. A total of 108 patients agreed to undergo the screening, and forty-seven patients were confirmed to have metabolic syndrome. Patients with metabolic syndrome or BMIs > 25 kg/m2 were invited to participate in the research. In total, sixty-two patients satisfied the inclusion criteria, and 22 patients consented to participate in the experiment.

Each participant was assigned one number from 1 to 22 by the first author. The second author enrolled participants. They were randomized to either Baduanjin program group or routine care group in a 1:1 ratio using blocked randomization having a block size of 4 by the fourth author. Patients in the experimental group (EG) participated in the Baduanjin intervention in a privacy setting", which involved 60-min sessions 3 times per week, 1 h after dinner between 6 and 7 pm; the entire program continued for 12 weeks. The control group (CG) received routine care and was required to walk during 6-7 pm. The outcome indicators for this intervention program involved the risk factors for metabolic syndrome, BW, and BMI.

When schizophrenia becomes chronic, patients experience lack of motivation. This exercise program aimed to increase patient participation and control their BW through Baduanjin program. The entire program continued for 3 months (mid-September to mid-December 2014), and the intervention was performed for 60 min 3 times per week; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program. While these participants practiced the Baduanjin program, the CG participants walked for 15-20 min in their wards.

ELIGIBILITY:
Inclusion Criteria:

* People were diagnosed with schizophrenia at the age of 20-65 years.
* People had taken regular antipsychotic medication for more than 10 weeks
* People lacked regular exercise in the past 3 months.
* People consented to receive blood collection and complete a questionnaire.
* People satisfied the modified Adult Treatment Panel III criteria for Asians i.e., three abnormal results for metabolic syndrome or two abnormal results with BMI > 25)

Exclusion Criteria:

* People with organic mental disorders, alcohol dependence, and substance abuse.
* people who are not willing to sign the consent.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Body weight | 3 months
  Change from Baseline Body weight (kilograms) at 3 months
body Mass Index (BMI). | 3 months
  BMI is defined as Body weight(kilograms) divided by height (meter) squared

SECONDARY OUTCOMES:
Fasting blood sugar | 3 months
  Change from Baseline Fasting blood sugar (mg/dl) at 3 months
Waist circumference | 3 months
  Change from Baseline Waist circumference (inches) at 3 months
triglyceride | 3 months
  Change from Baseline triglyceride (mg/dl) at 3 months
Blood pressure | 3 months
  Change from Baseline Blood pressure (mmHg) at 3 months
high-density lipoprotein | 3 months
  Change from Baseline high-density lipoprotein (mg/dl) at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Yueh Yang, Principal Investigator — ICMJE